CLINICAL TRIAL: NCT00471484
Title: A Phase II Trial of Oxaliplatin/Adriamycin/5 Fluorouracil in Continuous Infusion / Interferon α-2b (OXAFI) Combination as Neoadjuvant Therapy in Unresectable Non-Metastatic Hepatocellular Carcinoma
Brief Title: Combination Chemotherapy and Interferon Alfa-2b in Treating Patients With Nonmetastatic Liver Cancer That Cannot Be Removed by Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Centre, Singapore (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000543536; SINGAPORE-OC-GI-01-06; SINGAPORE-IRB-06-16-HEP; SINGAPORE-CTC0600327; SPRI-SINGAPORE-OC-GI-01-06
Record Dates: First submitted 2007-05-08; First posted 2007-05-10 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2008-11

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; localized unresectable adult primary liver cancer; advanced adult primary liver cancer; childhood hepatocellular carcinoma; stage III childhood liver cancer; stage IV childhood liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Introns; Doxorubicin; Fluorouracil; Oxaliplatin; Immunoenzyme Techniques; Immunohistochemistry; Chemotherapy, Adjuvant; Biopsy; Neoadjuvant Therapy

INTERVENTIONS:
Biological: recombinant interferon alfa-2b
Drug: doxorubicin hydrochloride
Drug: fluorouracil
Drug: oxaliplatin
Other: diagnostic laboratory biomarker analysis
Other: immunoenzyme technique
Other: immunohistochemistry staining method
Procedure: adjuvant therapy
Procedure: biopsy
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as oxaliplatin, doxorubicin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Interferon alfa may interfere with the growth of tumor cells. Giving combination chemotherapy together with interferon alfa may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with interferon alfa-2b works in treating patients with nonmetastatic liver cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with unresectable, nonmetastatic hepatocellular carcinoma treated with neoadjuvant oxaliplatin, doxorubicin hydrochloride, fluorouracil, and recombinant interferon alfa-2b.

Secondary

* Determine the overall survival of patients treated with this regimen.
* Determine the progression-free survival of patients treated with this regimen.
* Determine the rate of conversion to resectability of tumor in patients treated with this regimen.
* Determine the toxicity profile of this regimen in these patients.
* Assess the quality of life of patients treated with this regimen.
* Correlate changes in serological markers of angiogenesis before and after treatment with clinical outcome in these patients.
* Correlate and validate the use of functional imaging before and after treatment with clinical outcome in these patients.

OUTLINE: Patients receive neoadjuvant OXAFI therapy comprising oxaliplatin IV and doxorubicin hydrochloride IV on days 1, 8 and 15; fluorouracil IV continuously on days 1-28; and recombinant interferon alfa-2b subcutaneously three times weekly in weeks 1-4. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients receive at least 2 courses of neoadjuvant therapy before undergoing evaluation for response. Patients whose disease becomes resectable after achieving a complete or partial response proceed to surgery. Patients whose disease remains unresectable are reevaluated until their disease either becomes resectable, they complete neoadjuvant therapy, or they meet discontinuation criteria.

At least 2 weeks after receiving neoadjuvant therapy, patients whose disease is resectable undergo surgery for potentially complete resection of their tumors with curative intent. Patients who achieve complete resection proceed to adjuvant therapy.

At least 4 weeks after surgery, patients may restart OXAFI as adjuvant therapy, provided they have fully recovered from surgery and have received fewer than 6 courses of neoadjuvant therapy. Adjuvant therapy repeats every 28 days for a total of 6 courses (including neoadjuvant OXAFI) in the absence of disease progression or unacceptable toxicity.

Patients undergo blood and tissue collection at baseline and periodically during study for evaluation of circulating and tissue biomarkers of angiogenesis. Serum from venous blood samples is analyzed for concentration of VEGF by ELISA. Tumor tissue obtained before and after treatment is examined for tumor VEGF expression, microvessel density, and cellular proliferation by IHC.

Patients complete quality of life questionnaires at baseline, monthly during study treatment, after course 6 of neoadjuvant chemotherapy, or upon discontinuation of study treatment.

Patients are followed periodically for up to 5 years after curative resection of their tumors.

PROJECTED ACCRUAL: A total of 54 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed hepatocellular carcinoma

  * Advanced, unresectable, nonmetastatic disease
  * Multifocal disease within the same lobe of the liver allowed
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
* No intractable ascites that cannot be controlled by medical therapy
* No extrahepatic metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy > 3 months
* WBC ≥ 3,000/mm³
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Bilirubin ≤ 2.9 mg/dL
* AST and ALT ≤ 5 times upper reference range (URR)
* Albumin > 30 g/L
* Creatinine ≤ 1.5 times URR
* Creatinine clearance > 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study therapy
* No other prior malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No concurrent substantial medical illness, such as cardiac or renal disease
* MUGA heart study normal
* No history of allergic reactions attributed to compounds of similar chemical or biological composition used in the study
* No history of autoimmune disease
* No thyroid dysfunction
* No active hepatitis B or C flare or chronic active hepatitis
* Hepatitis B surface antigen (HBsAg) status known

  * If HBsAg is negative, anti-HBc antibodies should be tested; if anti-HBc is positive, then hepatitis B virus (HBV) DNA detection should be performed to discern presence of mutant HBV carriage
* No alcohol or drug abuse
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
* No psychiatric illness or social situation that would preclude study compliance

  * Patients with a history of depression or psychiatric disorders are ineligible

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy and/or radiotherapy
* No other concurrent investigational agents

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2007-03

PRIMARY OUTCOMES:
Objective tumor response rate as measured by RECIST criteria

SECONDARY OUTCOMES:
Serum VEGF levels
Tissue VEGF expression

CONTACTS AND LOCATIONS:
Overall Officials: Donald Poon, MD, Study Chair — National Cancer Centre, Singapore; Kian Fong Foo, MD — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre - Singapore, Singapore, Singapore

REFERENCES:
- [Result] Ang MK, Poon D, Foo KF, Chung YF, Chow P, Wan WK, Thng CH, Ooi L. A new chemoimmunotherapy regimen (OXAFI) for advanced hepatocellular carcinoma. Hematol Oncol Stem Cell Ther. 2008 Jul-Sep;1(3):159-65. doi: 10.1016/s1658-3876(08)50024-0. PMID 20063546